CLINICAL TRIAL: NCT05321199
Title: Efficacy of Intraoperative Use of Tranexamic Acid in Reducing Blood Loss During Telescoping Nail Application in Osteogenesis Imperfecta - Randomized Control Trials
Brief Title: Tranexamic Acid During Telescoping Nail Application In Osteogenesis Imperfecta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ammar Jamal Aldeen Mohammed Mohammed, Resident doctor, Assiut University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: TXA in OI
Record Dates: First submitted 2022-03-11; First posted 2022-04-11 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control patients (Experimental): Closed Envelope for group A (control); patients receiving no tranexamic acid. With Double-Blind Study in which the participants and observers are unaware of who receives tranexamic acid. The total blood loss (TBL), intraoperative blood loss (IBL), postoperative blood loss (PBL), hemoglobin (HGB) levels and Hematocrit value (Hct) on preoperatively (pre-op) and postoperatively, and amount of allogenic blood transfusion were recorded. Furthermore, the general information was also compared between groups.
  Interventions: Drug: Tranexamic acid
- Case patients (Experimental): Closed Envelope for group B (case); patients receiving tranexamic acid intravenously and topically. With Double-Blind Study in which the participants and observers are unaware of who receives tranexamic acid. The total blood loss (TBL), intraoperative blood loss (IBL), postoperative blood loss (PBL), hemoglobin (HGB) levels and Hematocrit value (Hct) on preoperatively (pre-op) and postoperatively, and amount of allogenic blood transfusion were recorded. Furthermore, the general information was also compared between groups.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic acid (TXA) is an antifibrinolytic drug that has been shown to be effective in reducing blood loss and the need for transfusions after several orthopaedic surgeries.
  Other Names: Kapron

SUMMARY:
The aim of this study is to assess the effective of intraoperative use of tranexamic acid in reducing blood loss during telescoping nail application in cases of osteogenesis imperfecta.

DETAILED DESCRIPTION:
Osteogenesis imperfecta (OI) is a rare inherited pathology that consists of abnormal type one collagen synthesis that affects all structures in the body. The most important and early sign of this pathology is the appearance of fractures after low-energy trauma, progressive bowing of long bones, joint instability, and chronic bone pain. The most used classification is the one created by Sillence that initially had four types and now is expended to more than 15 types. A new nomenclature was published in 2014 in order to simplify the classification and help understand such an intricate pathology. Clinically, all systems in the body are affected, but changes to the musculoskeletal are the most severe; besides, a variable degree of bone brittleness is present. Patients are suffering from severe hyperlaxity, short stature, scoliosis, progressive bowing of the limbs, and chronic bone pain due to continuous microfractures.

The surgical treatment of osteogenesis imperfecta (OI) is negatively influenced by clinical features such as osteoporosis, limb deformities and bone changes caused by bisphosphonate therapy. Blood loss during telescoping nail application in patients with Osteogenesis Imperfecta is a serious problem especially patients with Osteogenesis Imperfecta type III are considered at high risk of blood loss during surgery because of capillary fragility and an altered platelet function.

Tranexamic acid (TXA) is an antifibrinolytic drug that has been shown to be effective in reducing blood loss and the need for transfusions after several orthopaedic surgeries.

However, the effectiveness of tranexamic acid use in application of telescoping nail in osteogenesis imperfecta still remains unclear and no previously available study about this subject. The purpose of this study is to assess the effectiveness of intraoperative use of intravenous (IV) tranexamic acid in reducing total blood loss and transfusion rates for patients who will be operated with telescoping nail application for osteogenesis imperfecta.

Each patient with osteogenesis imperfecta, who consecutively will undergo telescoping femoral nail application with intraoperative use of tranexamic acid during 2022-2023, will be recruited in the study.

A total of 40 patients undergoing telescoping femoral nail application for osteogenesis imperfecta will be including in a prospective randomized study.

Taking detailed history and full clinical examination to exclude the presence of any medical disorder that prevents use of Tranexamic acid. Preoperative lab investigations are Complete Blood Count (CBC) to determine Hemoglobin HB level and Hematocrit value preoperatively.

Operations will be performing under general anesthesia, no tourniquet is using, and the intraoperative regime will be the same for all patients. Patients will be dividing into 2 groups; in group A (control); patients receiving no tranexamic acid, in group B (case); patients receiving 10-15mg/kg or 1g of tranexamic acid intravenously, given 30 minutes before skin incision in telescoping femoral nail application followed by another dose of intravenous tranexamic acid (10-15mg/kg; body weight average 1g) at time of wound closure.

Intraoperative blood loss shall be quantified by measuring irrigation fluid and the weight of surgical sponges used to dry the field intraoperatively by the researcher plus amount of blood in suction drain.

Comparison of blood loss between patients with first femoral osteotomy and patients with previous recurrent femoral osteotomies.

ELIGIBILITY:
Inclusion Criteria:

All patients with osteogenesis imperfecta who will undergo telescoping femoral nail application in Assiut University Hospital - Department of Orthopaedic and Trauma Surgery between April 2022 and March 2023.

Exclusion Criteria:

* Known allergy to Tranexamic Acid
* History of any acquired disturbances of colour vision
* History of major comorbidities (e.g., severe ischemic heart disease)
* Refusal of blood products
* History of fibrinolytic disorders requiring intraoperative antifibrinolytic treatment, coagulopathy in the past and/or as identified by a preoperative platelet count of <150,000/mm3, or a prolonged partial thromboplastin time, active intravascular clotting & known congenital thrombophilia
* Preoperative use of anticoagulant therapy within five days before surgery
* Medical Unfit
* Participation in another clinical trial involving pharmaceutical drugs.
* Patients or their relatives who refuse to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of change in mean blood loss in tranexamic acid group. | Baseline
  Based on determining the main outcome variable, the estimated minimum required sample size is 40 patients (20 in each group).
  The sample size was calculated using G*power software 3.1.9.2., based on the following assumptions:
  Main outcome variable is intraoperative blood loss in cases of Osteogenesis Imperfecta undergoing telescoping nail application which receive tranexamic acid vs. not received it.
  Main statistical test is one sided t-test to detect the difference between the two groups.
  Alpha = 0.05, Power = 0.80, Effect size = 0.81, Allocation ratio= 1

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Elbaseet, Lecturer, Study Director — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

REFERENCES:
- [Background] Sillence DO, Senn A, Danks DM. Genetic heterogeneity in osteogenesis imperfecta. J Med Genet. 1979 Apr;16(2):101-16. doi: 10.1136/jmg.16.2.101. PMID 458828
- [Background] Forlino A, Cabral WA, Barnes AM, Marini JC. New perspectives on osteogenesis imperfecta. Nat Rev Endocrinol. 2011 Jun 14;7(9):540-57. doi: 10.1038/nrendo.2011.81. PMID 21670757
- [Background] Van Dijk FS, Sillence DO. Osteogenesis imperfecta: clinical diagnosis, nomenclature and severity assessment. Am J Med Genet A. 2014 Jun;164A(6):1470-81. doi: 10.1002/ajmg.a.36545. Epub 2014 Apr 8. PMID 24715559
- [Background] Palomo T, Fassier F, Ouellet J, Sato A, Montpetit K, Glorieux FH, Rauch F. Intravenous Bisphosphonate Therapy of Young Children With Osteogenesis Imperfecta: Skeletal Findings During Follow Up Throughout the Growing Years. J Bone Miner Res. 2015 Dec;30(12):2150-7. doi: 10.1002/jbmr.2567. Epub 2015 Jun 30. PMID 26059976
- [Background] Thomas IH, DiMeglio LA. Advances in the Classification and Treatment of Osteogenesis Imperfecta. Curr Osteoporos Rep. 2016 Feb;14(1):1-9. doi: 10.1007/s11914-016-0299-y. PMID 26861807
- [Background] Hathaway WE, Solomons CC, Ott JE. Platelet function and pyrophosphates in osteogenesis imperfecta. Blood. 1972 Apr;39(4):500-9. No abstract available. PMID 4334923
- [Background] Armstrong D, VanWormer D, Solomons CC. Increased inorganic serum pyrophosphate in serum and urine of patients with osteogenesis imperfecta. Clin Chem. 1975 Jan;21(1):104-8. No abstract available. PMID 163711
- [Background] Russell RG, Bisaz S, Donath A, Morgan DB, Fleisch H. Inorganic pyrophosphate in plasma in normal persons and in patients with hypophosphatasia, osteogenesis imperfecta, and other disorders of bone. J Clin Invest. 1971 May;50(5):961-9. doi: 10.1172/JCI106589. PMID 4324072
- [Background] Jennings JD, Solarz MK, Haydel C. Application of Tranexamic Acid in Trauma and Orthopedic Surgery. Orthop Clin North Am. 2016 Jan;47(1):137-43. doi: 10.1016/j.ocl.2015.08.014. PMID 26614928
- [Background] Faraoni D, Goobie SM. The efficacy of antifibrinolytic drugs in children undergoing noncardiac surgery: a systematic review of the literature. Anesth Analg. 2014 Mar;118(3):628-36. doi: 10.1213/ANE.0000000000000080. PMID 24557107